CLINICAL TRIAL: NCT00283998
Title: Phase 4 Study Comparing Surigcal to Conservative Management of Type 2 Odontoid Fractures
Brief Title: Comparing Surgical to Conservative Management in the Treatment of Type II Odontoid Fractures Among the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: AOSpine North America (Industry)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-Odont-02
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Odontoid Fractures Type II
Keywords: Odontoid; Type II fractures; Elderly patients; Surgical vs. conservative treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: surgical versus conservative treatment — Surgical treatment of fractures versus conservative stabilization

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of surgical versus conservative management of type II odontoid fractures among patients >/= 65 years of age. Of secondary interest is to determine if there are differences in outcomes between anterior screw fixation and posterior fusion of these fractures.

ELIGIBILITY:
Inclusion Criteria:

* All new type II odontoid fractures including < those in which the fracture line crosses into the body of C2 < as long as it doesn't enter the superior articular process of C2
* Age 65+
* Stable and unstable fractures
* < 3 months postinjury
* No previous treatment for an odontoid fracture

Exclusion Criteria:

* Pathologic fractures unrelated to osteoporosis
* Severe dementia or other severe mental health problem if there is no consentable surrogate available
* Participating in other trials or unlikely to attend follow-ups

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Quality of life using the Neck disability Index | 12 months
Quality of life using the SF-36 | 12 months
Proportion of bony fusion between the two treatments | 6 months
Proportion rate of non-union between the two treatments | 6 months

SECONDARY OUTCOMES:
Rate of complications | 12 months
Cervical range of motion | 12 months
Identify the risk factors for a poor outcome independent of treatment intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Vaccaro, MD, Principal Investigator — Th. Jefferson University Philadelphia
Locations (1):
- Emory University SOM: Orthopedics, Atlanta, Georgia, United States